CLINICAL TRIAL: NCT03580304
Title: Evaluation of Mental and Physical Load During Lab-simulated Industrial Work
Brief Title: Evaluation of Physical and Cognitive Industrial Workload
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Romain Meeusen, Prof. Dr., Vrije Universiteit Brussel
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: S008517N
Record Dates: First submitted 2018-05-11; First posted 2018-07-09 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Work-Related Condition; Physical Stress; Mental Fatigue
Keywords: Fatigue Mental; Fatigue Signs and Symptoms; Behavioral Symptoms; Industrial work; physical effort; mental effort; questionnaires; ergonomic evaluation
MeSH Terms: conditions — Mental Fatigue; Behavioral Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- industrial-physical-cognitive (Experimental)
  Interventions: Behavioral: Industrial work; Behavioral: Physical load; Behavioral: Cognitive load
- industrial- cognitive-physical (Experimental)
  Interventions: Behavioral: Industrial work; Behavioral: Physical load; Behavioral: Cognitive load
- physical- industrial- cognitive (Experimental)
  Interventions: Behavioral: Industrial work; Behavioral: Physical load; Behavioral: Cognitive load
- physical-cognitive- industrial (Experimental)
  Interventions: Behavioral: Industrial work; Behavioral: Physical load; Behavioral: Cognitive load
- cognitive- industrial-physical (Experimental)
  Interventions: Behavioral: Industrial work; Behavioral: Physical load; Behavioral: Cognitive load
- cognitive-physical-industrial (Experimental)
  Interventions: Behavioral: Industrial work; Behavioral: Physical load; Behavioral: Cognitive load

INTERVENTIONS:
Behavioral: Industrial work — Subjects perform simulated industrial work in lab setting. The industrial task exists of a physical component and a cognitive component. Physical load is measured by questionnaires and basic physiological measurements (e.g. heart rate). Mental fatigue will be determined by questionnaires and a cognitive stroop task before and after the trial.
Behavioral: Physical load — The physical load of an industrial task will be simulated during this intervention. Physical load is measured by questionnaires and basic physiological measurements (e.g. heart rate). Before and after the trial, mental fatigue will be determined by questionnaires and a cognitive stroop task (10 min)
Behavioral: Cognitive load — The cognitive load of an industrial task will be simulated in this intervention. Physical load is measured by questionnaires and basic physiological measurements (e.g. heart rate). Before and after the trial, mental fatigue will be determined by questionnaires and a cognitive stroop task (10 min)

SUMMARY:
The main aim of the project is to evaluate a novel upper body exoskeleton during simulated industrial work. In this stage of the project, a study analysing the physical and mental load during occupational work will be carried out. High risk tasks will be identified in the field and simulated in lab-setting to analyse physical and mental load using physiological and biomechanical data.These will include, but will not be limited to, non-ergonomic postures, for example performing operations above the head or reaching in front of, to the side of, or behind the body; flexing the arms for extended periods of time; and bending or twisting the torso to lift an object from low or distant locations. Important items to assess in this task are the frequency and duration of tasks and activities, lifting characteristics, perceived physical effort and work-induced fatigue.

ELIGIBILITY:
Inclusion Criteria:

* male
* 18 - 65 yrs old

Exclusion Criteria:

* injury

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
EEG: change in power spectral density (change in mental fatigue: physiological component) | Measuring EEG during Stroop tasks (10 minutes) before and after each 90 minute task
  The power of different frequency bands during a cognitive Stroop task will be compared PRE vs POST 90 minute task and differences between different tasks will be analysed.

SECONDARY OUTCOMES:
EEG: changes in event related potentials during cognitive Stroop task (change in mental fatigue: physiological component) | Measuring EEG during Stroop tasks (10 minutes) before and after each 90 minute task
  Event related potentials during cognitive Stroop task will be compared PRE vs POST 90 minute task and differences between different tasks will be analysed.
Change in mental fatigue (behavioral component: part 1) | Measuring reaction time during Stroop tasks (10 minutes) before and after each 90 minute task
  Reaction time during cognitive stroop task
Change in mental fatigue (behavioral component: part 2) | Measuring accuracy during Stroop tasks (10 minutes) before and after each 90 minute task
  Accuracy time during cognitive stroop task
Change in mental fatigue (subjective component) | Before and after each 90 minute task subjective questionnaire will be filled out
  Questionnaire (sRPE) before and after performing each 90 min task

CONTACTS AND LOCATIONS:
Overall Officials: Romain Meeusen, Prof. Dr., Principal Investigator — Vrije Universiteit Brussel
Locations (1):
- Lichamelijk Opvoeding en Kinesitherapie, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-11): https://cdn.clinicaltrials.gov/large-docs/04/NCT03580304/Prot_SAP_000.pdf